CLINICAL TRIAL: NCT00968552
Title: Prospective Evaluation of the Clinical Utility of Endoscopically Placed Self-expandable Stents
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: Stents/ERCP
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Gastrointestinal Diseases
Keywords: Any Gastrointestinal problem that would require an endoscopically placed stent
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing stent placement: Patients who are scheduled to undergo stent placement via endoscopy as part of their routine medical care.
  Interventions: Procedure: Self-expandable stent placement via endoscopy

INTERVENTIONS:
Procedure: Self-expandable stent placement via endoscopy — Self-expandable stent placement via endoscopy

SUMMARY:
The investigators' believe that it is important to medical practice to obtain information on how expandable metal stents work in a large group of patients who have metal stents placed in the gastrointestinal system. The purpose of this research study is to collect information on the stent placement in our facility and how the patients responded to the stent placement.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Scheduled to undergo endoscopy with placement of self-expanding stent at the University of Florida, Gainesville, FL.
3. Subject must be able to give informed consent.

Exclusion Criteria:

1. Any contraindication to performing endoscopy.
2. Participation in another research protocol that could interfere or influence the outcomes measures of the present study.
3. The subject is unable/unwilling to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Age 18 or older
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2009-08; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
The purpose of this research study is to collect information on the stent placement in our facility and how the patients responded to the stent placement. | at the time of stent placement

CONTACTS AND LOCATIONS:
Locations (1):
- Shands UF endoscopy Center, Gainesville, Florida, United States

REFERENCES:
- [Derived] Wagh MS, Draganov PV. Per-oral endoscopic tunneling for restoration of the esophagus: a novel endoscopic submucosal dissection technique for therapy of complete esophageal obstruction. Gastrointest Endosc. 2017 Apr;85(4):722-727. doi: 10.1016/j.gie.2016.08.035. Epub 2016 Sep 7. PMID 27612924